CLINICAL TRIAL: NCT04503720
Title: Continuous Local Anaesthetic Wound Infusion (CLoWI) Versus PCA Morphine for Pain Control After Major Abdominal Surgery:A Double Blinded, Randomized, Controlled, Non Inferiority Trial (CLoWI Trial)
Brief Title: CLoWI Versus PCA Morphine for Pain Control After Major Abdominal Surgery
Acronym: CLoWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JurongHealth (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Juronghealth
Record Dates: First submitted 2020-02-26; First posted 2020-08-07 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Surgical Wound; Post-Op Complication; Opioid Use
Keywords: continuous local wound infusion; opioids; post-operative pain; surgical incision
MeSH Terms: conditions — Surgical Wound; Postoperative Complications; Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLoWI (Experimental): CLoWI (ropivacaine) and PCA (normal saline)
  The local anaesthetic infusion will be administered via 2 catheters using a ON-Q® (Halyard) delivery system that will be placed under direct vision by the surgeon at the time of wound closure. 40 mls of 0.25% ropivacaine are infiltrated in the preperitoneal plane. 0.5% ropivacaine will be infused at a rate of 4mls/hour (2mls/hour in each catheter).
  The dosage 40 mls of 0.25% ropivacaine and 0.5% ropivacaine at 4mls/hr (20mg/hr) over 4 days will be less than the recommended toxic dose of 3-4 mg/kg.
  Interventions: Device: CLoWI
- PCA (Active Comparator): PCA (Morphine) and CLoWI (normal saline)
  Morphine will be administered via the standard PCA protocol in accordance to the hospital's Acute Pain Service Programme:
  * Concentration: 1mg/ml
  * Bolus (Loading): 1mg
  * Lockout Interval: 5 minutes
  * Maximum hourly dose of 10mg
  Interventions: Device: PCA

INTERVENTIONS:
Device: CLoWI — Patients will receive a continuous wound infusion with ropivacaine and normal saline in the PCA pump.
  Arms: CLoWI
Device: PCA — Patients will receive a continuous wound infusion with normal saline and morphine in the PCA pump.
  Arms: PCA

SUMMARY:
Major abdominal surgery is associated with significant complications which may lead to morbidity and mortality. Pain experienced after surgery affects the recovery from surgery.

Our study aims to evaluate the current gold standard of PCA morphine infusion against a continuous wound infusion (CLoWI). The use of CLoWI negates the side-effects of opioids, and will be the first randomised controlled trial to compare PCA (Morphine) with CLoWI-LA (Ropivacaine).

DETAILED DESCRIPTION:
Major intra-abdominal surgery represents one of the commonest groups of surgical procedures performed both worldwide and within Singapore. Common general surgical conditions requiring major intra-abdominal surgery include intestinal pathologies such as cancer, ischaemia, infection, haemorrhage and perforation.

Major surgery within the abdominal cavity is associated with significant complications which may be life threatening with an associated hospital mortality rate of as high as 20% for emergency surgery. Importantly, the recovery from this type of major surgery often entails significant pain and discomfort for the patient during healing of the abdominal wound and internal organs from tissue trauma associated with these surgical procedures.

Recent developments in major intra-abdominal surgery have demonstrated the importance of the early surgical recovery period where common postoperative complications including pain, chest infection, intestinal ileus and delerium are not only associated with prolonged hospital stay but are harbingers of poor long term surgical outcomes. Current recommendations for perioperative management of patients undergoing major intra-abdominal surgery stress the importance of high quality perioperative care to minimise these sequelae. Key features of these recommendations are to provide a pain free postoperative surgical recovery with minimal nausea and vomiting to facilitate early mobilisation and functional recovery from surgery.

Patient controlled analgesia (PCA) with opioids is the first line analgesia therapy currently used in the immediate post-operative period following major abdominal surgery. PCA with opioids has some inherent disadvantages that include side-effects of opioids such as nausea, vomiting, prolonged ileus, dizziness, hallucination and respiratory depression with the need for supplementary oxygen. This is most pertinent in elderly patients who are more prone to these side-effects in addition to being more likely to have difficulties in understanding how to use the PCA and so are more vulnerable to inadequate pain control. Consequently, there may be a delay in resuming mobility and discharge from hospital.

Continuous local wound infusion (CLoWI) with Ropivacaine that is delivered into the extraperitoneal plane via an ON-Q® (Halyard) infusion pump has been shown to be an effective analgesia post-operatively. The use of CLoWI negates the side-effects of opioids and furthermore, the small portable pump allows early ambulation with no requirement for supplementary oxygen. Previous published research has demonstrated the benefits of continuous local wound infusion with local anaesthesia in terms of postoperative analgesia and surgical recovery However, there are no randomized controlled trials comparing PCA versus continuous local wound infusion alone; this study will be the first randomised controlled trial to compare PCA (Morphine) with CLoWI-LA (Ropivacaine).

The local anaesthetic drug to be used for the wound infiltration system is Ropivacaine. Its mechanism of action involves inhibiting sodium influx through sodium-specific ion channels in the peripheral nerve axonal cell membrane, in particular, the voltage gated sodium channels. When the influx of sodium is interrupted, an action potential cannot arise and the conduction of a pain signal is inhibited. The local anaesthetic will be administered via 2 catheters that will be placed under direct vision by the surgeon at the time of wound closure.

Ropivacaine 0.5% will be infused at a rate of 4mls/hour (2mls/hour in each catheter) for a total of 4 days. It is currently in clinical use within our hospital as a routine method of providing postoperative analgesia following major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective or urgent# open abdominal surgery

Abdominal Surgery may include the following procedures:

A) Urgent laparotomy for perforated viscus, intestinal obstruction. B) Elective abdominal surgery for upper and lower gastrointestinal surgery

* Ability to provide informed consent. A signed and dated written informed consent prior to study participation.
* Age 21 to 80 years for both males and females

Exclusion Criteria:

* Female subject who is pregnant
* Inability to comply with PCA instructions due to physical disabilities. For example, visual or hearing impairment, arthritis, peripheral neuropathy.
* Known allergy to local anaesthetic or opioid drugs (Morphine).
* Current or recent on opioid therapy. For example due to chronic pain illness, opioid (or other) drug abuse or recent surgery.
* Severe comorbid diseases including liver cirrhosis, renal failure requiring dialysis, Grade 4 NYHA (New Yoke Heart Association) heart failure, respiratory illness requiring NIV (Non-Invasive Ventilation), etc.
* Severe associated acute illness American Society of Anesthesiologists (ASA) Grade 4 or 5 where survival following surgery is not expected

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To compare CLoWI and PCA (Morphine) in terms of post operative pain control | 5 days
  To determine if wither CLoWI or PCA will achieve better post-operative pain control based on a numerical rating score from 0 - 10

SECONDARY OUTCOMES:
To compare CLoWI and PCA (Morphine) in terms of post operative complication rates associated with opioid usage | 5 days
  This includes the following complications - urinary retention, time to flatus, time to bowel opening, nausea and vomiting.
To compare CLoWI and PCA (Morphine) in terms of the length of postoperative hospital stay. | from the time of surgery till discharge, an average of 5 days
  This takes into account the length of time the patient spends in the hospital between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Keh, FRCS, Principal Investigator — Ng Teng Fong General Hospital
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang SS, Ying AJ, Affan ET, Kakala BF, Strippoli GF, Bullingham A, Currow H, Dunn DW, Yeh ZY. Continuous local anaesthetic wound infusion for postoperative pain after midline laparotomy for colorectal resection in adults. Cochrane Database Syst Rev. 2019 Oct 19;10(10):CD012310. doi: 10.1002/14651858.CD012310.pub2. PMID 31627242
- [Background] Prochazka V, Svoboda M, Svaton R, Grolich T, Farkasova M, Kala Z. Use of preperitoneal wound catheter for continuous local anaesthesia after laparoscopic colorectal surgery. Rozhl Chir. 2019 Summer;98(9):356-361. doi: 10.33699/PIS.2019.98.9.356-361. PMID 31698911
- [Background] Dalmau A, Fustran N, Camprubi I, Sanzol R, Redondo S, Ramos E, Torras J, Sabate A. Analgesia with continuous wound infusion of local anesthetic versus saline: Double-blind randomized, controlled trial in hepatectomy. Am J Surg. 2018 Jan;215(1):138-143. doi: 10.1016/j.amjsurg.2017.09.007. Epub 2017 Sep 20. PMID 28958651